CLINICAL TRIAL: NCT01595191
Title: Bach Music in Preterm Infants: No "Mozart Effect" on Resting Energy Expenditure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Principal Investigator, Michal Roll PhD,MBA, Head, Research institute, Tel-Aviv Sourasky Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 07-346 TLV
Record Dates: First submitted 2012-05-08; First posted 2012-05-09 (Estimated); Last update posted 2012-05-09 (Estimated); Status verified 2012-05

CONDITIONS: Resting Energy Expenditure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Music by Mozart (Active Comparator): The sequence by which Bach, Mozart, or no music were administered (over 3 consecutive days) was determined by randomization using random numbers. Infants listened to Bach or Mozart using the compact discs entitled "Baby Bach" and "Baby Mozart" (Baby smart, Nir Zvi, Israel). The music was played using a music player at a volume of 65-70 dB with attached speakers which were placed at a distance of 30 cm from the infant's ears. According to the American Academy of Pediatrics recommendations (5): the volume did not exceed 75dB and the background noise near the infant's ears was maintained below 45 dB. Music (Mozart or Bach) was initiated 10 minutes prior to the beginning of the metabolic measurements and continued for 30 minutes while energy expenditure (EE) was recorded. In the same manner EE was recorded for each infant with no music therapy.
  Interventions: Other: Mozart music
- Bach Music (Active Comparator): The sequence by which Bach, Mozart, or no music were administered (over 3 consecutive days) was determined by randomization using random numbers. Infants listened to Bach or Mozart using the compact discs entitled "Baby Bach" and "Baby Mozart" (Baby smart, Nir Zvi, Israel). The music was played using a music player at a volume of 65-70 dB with attached speakers which were placed at a distance of 30 cm from the infant's ears. According to the American Academy of Pediatrics recommendations (5): the volume did not exceed 75dB and the background noise near the infant's ears was maintained below 45 dB. Music (Mozart or Bach) was initiated 10 minutes prior to the beginning of the metabolic measurements and continued for 30 minutes while energy expenditure (EE) was recorded. In the same manner EE was recorded for each infant with no music therapy.
  Interventions: Other: Bach music

INTERVENTIONS:
Other: Bach music — Infants listened to Bach or Mozart using the compact discs entitled "Baby Bach" and "Baby Mozart" (Baby smart, Nir Zvi, Israel).
  Arms: Bach Music
Other: Mozart music — Infants listened to Bach or Mozart using the compact discs entitled "Baby Bach" and "Baby Mozart" (Baby smart, Nir Zvi, Israel).
  Arms: Music by Mozart

SUMMARY:
Exposure to Mozart music significantly lowers resting energy expenditure (REE) in healthy preterm infants. Whether this finding is related to music per-se or to music by Mozart is unknown. The objective is to study whether J.S. Bach music has a lowering effect on REE similar to that of Mozart music.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants at post menstrual age of 30-37 weeks who were appropriate for gestational age, clinically and thermally stable, gavage-fed, were eligible for recruitment.
* At the time of the study they were all tolerating full enteral feeding (150-160 cc/kg weight/day) without significant gastric residuals (<5% of total feed), they were all growing steadily, and had no electrolyte imbalance.
* All infants who were recruited successfully passed a hearing screening test prior to discharge (otoacoustic emission and automated auditory brainstem response)

Exclusion Criteria:

* Infants with significant complications of prematurity such as intraventricular hemorrhage, periventricular leucomalacia, necrotizing enterocolitis, active apneas of prematurity, patent ductus arteriosus, active infection, electrolyte imbalance and major congenital anomalies.

Ages: 5 Days to 59 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2010-07; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Resting energy expenditure | 3 CONSECUTIVE DAYS
  Metabolic measurements were performed by indirect calorimetry using the Deltatrac II Metabolic monitor (DateOhmeda, Helsinki, Finland). This system consists of a hood, which is placed over the infant's head and of two sensors. It uses the principle of an open circuit which allows for continuous measurements of O2 consumption and C02 production. The energy expenditure is calculated using the equation 5.5VO2+1.76VCO2.

CONTACTS AND LOCATIONS:
Overall Officials: Dror Mandel, MD, Principal Investigator — Direcrotr, NICU
Locations (1):
- Tel Aviv Medical Center, Tel Aviv, Israel

REFERENCES:
- [Background] Lubetzky R, Mimouni FB, Dollberg S, Reifen R, Ashbel G, Mandel D. Effect of music by Mozart on energy expenditure in growing preterm infants. Pediatrics. 2010 Jan;125(1):e24-8. doi: 10.1542/peds.2009-0990. Epub 2009 Dec 7. PMID 19969615